CLINICAL TRIAL: NCT00492492
Title: Treatement of Extension Fractures of the Distal Radius : Prospective Randomized Postoperative Comparison Between Trans-styloid and Intrafical Pinning on the One Side and Volar Fixed-angle Plating on the Other Side.
Brief Title: Treatement of Extension Fractures of the Distal Radius
Acronym: fradius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I06029
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Fracture of Distal Radius
Keywords: radius,; pinning,; fixed-angle plate,; quick-DASH,; HERZBERG-score.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trans-styloid and intrafocal pinning on the one side (Other): trans-styloid and intrafocal pinning on the one side
  Interventions: Procedure: trans-styloid and intrafocal pinning on the one side
- volar fixed-angle plating on the other side (Other): volar fixed-angle plating on the other side
  Interventions: Procedure: volar fixed-angle plating on the other side

INTERVENTIONS:
Procedure: trans-styloid and intrafocal pinning on the one side
  Arms: trans-styloid and intrafocal pinning on the one side
Procedure: volar fixed-angle plating on the other side
  Arms: volar fixed-angle plating on the other side

SUMMARY:
Treatment of extension fractures of the distal radius : prospective randomized postoperative comparison between trans-styloid and intrafocal pinning on the one side and volar fixed-angle plating on the other side.

DETAILED DESCRIPTION:
Distal radius fractures are more and more numerous. Most of the time, the people concerned are elderly or old with an osteoporotic bone, and an important dorsal metaphysal comminution. The French reference treatment of the extension distal radius fracture, the Kapandji method, turns out to be less and less performing to treat such complicated fractures. At the moment, two points of view are in opposition in France. On the one side, the point of view of those who are in favour of the treatment by intrafocal pinning: they think they will be able to improve their technique if they add a trans-styloid pinning of stabilisation. On the other side, those who are in favour of a treatment using a volar fixed-angle plating.

The purpose of the study is to compare these two types of treatment by using a prospective and randomized analysis.

The main judging criterion will lay on an X-ray assessment of the distal radius, we will try to find a loss of reduction at tree month.

The secondary criteria will lay on fonctional scores (quickDASH and Herzberg score) at 6 weeks, 3 months and 6 months, as well as on post-operative X-ray assessments in order to compare post-operative reduction of the distal radius fracture.

All the patients taken to the emergency ward of Limoges Hospital, and suffering from an extension distal radius fracture (intra or extra articular according to Kapandji classification) will have the possibility to participate in this study, if they want to.

The patients will be X-rayed before and after the operation, they will have an immobilization for 3 weeks. Then the cast will be removed, and new X-rays will be taken. Then the patients will be allowed to perform their daily activities. A new follow-up control will take place 6 week later, it will include a new series X-rays and functional scores. At this point, people will be able to start physiotherapy. New functional scores and X-ray assessments will still be taken 3 and 6 months later.

All the X-rays will be analyzed by an orthopaedist, a radiologist, and by a radiological software.

* Fonctional scores (quickDASH and Herzberg score) at 6 weeks, 3 months and 6 months.
* X-ray assessment after the operation and at 3 weeks, 6 weeks, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patient who is affiliated to the NHS (National Health Service)
* patient who has officially given his consent
* on over 50 year old patient
* Patient with an extension fracture of the distal radius
* patient who is in no condition to express his consent

Exclusion Criteria:

* patient who is under the protection of justice
* Patient with an open fracture
* Patient with an flexion fracture of the distal radius
* Patient with a metastasis localized in the distal radius
* traumatised patient
* patient who is liable not to profit by medical follow-up in Limoges hospital after he has been operated on
* A pregnant woman / a parturient / a breast-feeding mother
* patient who is serving a sentence .
* patient sent to hospital without his consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The main judging criterion will lay on an X-ray assessment of the distal radius, we will try to find a loss of reduction. | 3 months

SECONDARY OUTCOMES:
The secondary criteria will lay on fonctional scores (quickDASH and Herzberg score), as well as on post-operative X-ray assessments in order to compare post-operative reduction of the distal radius fracture. | 6 weeks, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis CHARISSOUX, MD, Principal Investigator — CHU LIMOGES
Locations (1):
- Department of Bone Surgery, Limoges, France

REFERENCES:
- [Background] Marcheix PS, Dotzis A, Benko PE, Siegler J, Arnaud JP, Charissoux JL. Extension fractures of the distal radius in patients older than 50: a prospective randomized study comparing fixation using mixed pins or a palmar fixed-angle plate. J Hand Surg Eur Vol. 2010 Oct;35(8):646-51. doi: 10.1177/1753193410364179. Epub 2010 Mar 17. PMID 20237186